CLINICAL TRIAL: NCT01560780
Title: Prasugrel for Prevention of Early Saphenous Vein Graft Thrombosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-007-11F
Record Dates: First submitted 2012-03-16; First posted 2012-03-22 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Bypass
Keywords: Coronary Artery Bypass; thrombosis; prasugrel
MeSH Terms: conditions — Thrombosis | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Prasugrel (Experimental): prasugrel 10 mg by mouth daily
  Interventions: Drug: Prasugrel
- Arm 2: Placebo (Placebo Comparator): placebo by mouth once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prasugrel — one 10 mg tablet by mouth daily
  Other Names: Effient
  Arms: Arm 1: Prasugrel
Drug: Placebo — placebo similar in appearance to prasugrel
  Arms: Arm 2: Placebo

SUMMARY:
This is a randomized-controlled clinical trial that will randomize 120 patients undergoing clinically-indicated coronary artery bypass graft surgery to prasugrel at a dose of 10 mg daily or matching placebo for 12 months, starting at the time of hospital dismissal from surgery. The primary goal of the study is to determine whether prasugrel administration will prevent thrombus (clot) formation within a saphenous vein graft at 12 months, as examined by optical coherence tomography.

DETAILED DESCRIPTION:
Aortocoronary saphenous vein graft failure is common and is associated with high morbidity and mortality. Thrombus formation plays a critical role in early saphenous vein graft occlusion and may predispose to subsequent atherosclerosis formation. Optical coherence tomography is a novel, high-resolution, intravascular imaging technique that can reliably identify thrombus. Based on the findings of earlier VA Cooperative Studies, aspirin significantly reduces the incidence of early saphenous vein graft failure and is currently used in nearly all patients undergoing coronary bypass graft surgery. Administration of clopidogrel for improving early saphenous vein graft patency has provided conflicting results in small randomized studies. Prasugrel is a novel thienopyridine that provides more rapid, consistent, and intense platelet inhibition than clopidogrel. However, in patients who undergo coronary artery bypass graft surgery, it remains unknown whether prasugrel may decrease thrombus formation in saphenous vein grafts during the first postoperative year, and whether this will result in less saphenous vein graft wall thickening, less lipid deposition in the saphenous vein graft wall and fewer clinical events without increasing the risk for severe bleeding.

Hypothesis: The investigators hypothesize that in patients undergoing clinically-indicated coronary artery bypass graft surgery, administration of prasugrel starting at dismissal from the index coronary bypass graft surgery hospitalization will result in lower prevalence of thrombus formation in a target SVG, as assessed by optical coherence tomography performed 12 months post surgery compared to placebo, with similar incidence of major bleeding.

This is a phase III, single-center, double-blind trial that will randomize 120 patients undergoing clinically-indicated coronary artery bypass graft surgery to prasugrel at a dose of 10 mg daily or matching placebo for 12 months, starting at the time of hospital dismissal from surgery. All patients will receive aspirin. Coronary angiography, optical coherence tomography, intravascular ultrasonography, and near-infrared spectroscopy of one target saphenous vein graft will be performed at 12 months to determine whether compared to placebo, administration of prasugrel will result in:

1. Reduction of the prevalence of intragraft thrombus at 12-month follow-up optical coherence tomography imaging (primary efficacy endpoint)
2. Similar incidence of severe bleeding using the Global Utilization of Streptokinase and t-PA for Occluded Coronary Arteries (GUSTO) criteria (primary safety endpoint)
3. Reduction in the incidence of angiographic SVG failure (defined as 75% SVG diameter stenosis in at least one SVG); reduction in total and normalized total target saphenous vein graft atheroma volume, as assessed by intravascular ultrasonography; and reduction of saphenous vein graft lipid core burden index, as assessed at near-infrared intracoronary spectroscopy at 12-month follow-up cardiac catheterization (secondary endpoints)
4. Reduction of major adverse cardiac events, defined as the composite of death, acute coronary syndrome, or coronary revascularization) during follow-up (secondary endpoints)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Willing and able to give informed consent. The patients must be able to comply with study procedures and follow-up.
* Undergoing clinically-indicated coronary artery bypass graft surgery

Exclusion Criteria:

* Known allergy to aspirin or prasugrel
* Need for concomitant cardiac procedure, such as valve repair or replacement
* Increased risk of bleeding, including need for warfarin or dabigatran administration
* Positive pregnancy test or breast-feeding
* Coexisting conditions that limit life expectancy to less than 12 months or that could affect a patient's compliance with the protocol
* Serum creatinine > 2.5 mg/dL
* Severe peripheral arterial disease limiting vascular access
* Prior stroke or transient ischemic attack
* Weight <60 kg or age >75 years
* Multiple distal SVG anastomoses
* Postoperative complications prolonging hospitalization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuaib M. Abdullah, MD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (4):
- United States (4):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Jesse Brown VA Medical Center Community-Based Outpatient Clinic Lake Side Divison, Chicago, IL, Chicago, Illinois
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
Started | 42 | 42
Clinical Follow-Up at 12 Months | 42 | 42
Completed Study Drug for 12 Months | 27 | 27
Completed (Underwent Angiography at 12 months) | 29 | 30
Not Completed | 13 | 12
Not completed — Death | 2 | 1
Not completed — Patient Preference | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 64 (6) | 64 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 41 | 41 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 31 | 32 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Intragraft Thrombus at 12-month Follow-up Optical Coherence Tomography Imaging
Description: Number of patients with intragraft thrombus seen at 12 month follow-up by optical coherence tomography in imaged saphenous vein graft
Time Frame: 12 months
Population: In the prasugrel arm, 29 of the 42 patients underwent SVG angiography at 12 months (2 died, 11 did not want to undergo SVG angiography). Of these, 25 had interpretable OCT.
  In the placebo arm, 30 of the 42 patients underwent SVG angiography at 12 months (1 died, 11 did not wish to undergo SVG angiography). Of these, 28 had interpretable OCT.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
Number analyzed (Participants) | 25 | 28
Participants | 14 | 14
Statistical Analysis 1: Comparison: Arm 1: Prasugrel vs Arm 2: Placebo; Test type: Superiority; p = 0.78, Fisher Exact

2. Secondary Outcome: Number of Patients With Severe Bleeding Using the Global Utilization of Streptokinase and t-PA for Occluded Coronary Arteries (GUSTO) Criteria
Description: Number of patients with major bleeding defined by the Global Utilization of Streptokinase and t-PA for Occluded Coronary Arteries criteria.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
Number analyzed (Participants) | 42 | 42
Participants | 1 | 0
Statistical Analysis 1: Comparison: Arm 1: Prasugrel vs Arm 2: Placebo; Test type: Equivalence — safety end-point with p-value of <0.05; p > 0.99, Log Rank

3. Secondary Outcome: Number of Patients With Angiographic Saphenous Vein Graft Failure
Description: Number of patients with angiographic saphenous vein graft failure (defined as =75% SVG diameter stenosis in at least one saphenous vein graft)
Time Frame: 12 months
Population: In the prasugrel arm, 29 of the 42 patients underwent SVG angiography at 12 months (2 died, 11 did not want to undergo SVG angiography).
  In the placebo arm, 30 of the 42 patients underwent SVG angiography at 12 months (1 died, 11 did not wish to undergo SVG angiography).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
Number analyzed (Participants) | 29 | 30
Participants | 7 | 12
Statistical Analysis 1: Comparison: Arm 1: Prasugrel vs Arm 2: Placebo; Test type: Superiority; p = 0.19, Fisher Exact

4. Secondary Outcome: Total Target Saphenous Vein Graft Atheroma Volume, as Assessed by Intravascular Ultrasonography
Description: Total target saphenous vein graft atheroma volume (mm3) as assessed by Intravascular ultrasound imaging in imaged saphenous vein grafts.
Time Frame: 12 months
Population: In the prasugrel arm, 29 of the 42 patients underwent SVG angiography at 12 months (2 died, 11 did not want to undergo SVG angiography). Of these, 25 had interpretable IVUS.
  In the placebo arm, 30 of the 42 patients underwent SVG angiography at 12 months (1 died, 11 did not wish to undergo SVG angiography). Of these, 27 had interpretable IVUS.
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
Number analyzed (Participants) | 25 | 27
mm3 | 349 (189) | 358 (175)
Statistical Analysis 1: Comparison: Arm 1: Prasugrel vs Arm 2: Placebo; Test type: Superiority; p = 0.85, t-test, 2 sided

5. Secondary Outcome: Saphenous Vein Graft Lipid Core Burden Index, as Assessed at Near-infrared Intracoronary Spectroscopy
Description: Lipid core burden as measured by Lipid Core Burden Index on near infrared intracoronary spectroscopy imaging of saphenous vein graft. Lipid Core Burden Index is defined as the fraction of pixels within the scanned region with a probability >0.60 that a lipid core plaque is present (calculated by an algorithm developed to identify the NIRS signals associated with the molecular structure of lipids), multiplied by 1000 using EchoPlaque software (INDEC Medical Systems; Los Altos, CA) . Thus, the lipid core burden index (LCBI) is a quantitative summary metric of the probability of the presence of lipid within the scanned region, with a range of 0-1000, with higher indices indicating a higher proportion of pixels with a >0.6 probability of lipid being present in the pullback of the catheter along the length of the entire vessel.
Time Frame: 12 months
Population: In the prasugrel arm, 29 of the 42 patients underwent SVG angiography at 12 months (2 died, 11 did not want to undergo SVG angiography). Of these, 12 had interpretable NIRS.
  In the placebo arm, 30 of the 42 patients underwent SVG angiography at 12 months (1 died, 11 did not wish to undergo SVG angiography). Of these, 20 had interpretable NIRS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
Number analyzed (Participants) | 13 | 20
units on a scale | 7.5 (9.3) | 7.4 (15.5)
Statistical Analysis 1: Comparison: Arm 1: Prasugrel; Test type: Superiority; p = 0.97, t-test, 2 sided

6. Secondary Outcome: Major Adverse Cardiac Events, Defined as the Composite of Death, Acute Coronary Syndrome, or Coronary Revascularization) During Follow-up
Description: Number of patients with the composite outcome of death, acute coronary syndrome, or coronary revascularization.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
Number analyzed (Participants) | 42 | 42
Participants | 8 | 4

7. Secondary Outcome: Normalized Total Target Saphenous Vein Graft Atheroma Volume, as Assessed by Intravascular Ultrasonography
Description: On IVUS images, atheroma volume was defined as the sum of the cross-sectional areas between the leading edges of the lumen and external elastic membrane. Total Target SVG atheroma volume was calculated as:
  ∑(EEM area - Lumen area).
  Normalized atheroma volume represents the atheroma volume corrected for pullback length, and this parameter was calculated as:
  ∑(EEM area - Lumen area)/number of frames in pullback
Time Frame: 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm3/frame
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
Number analyzed (Participants) | 25 | 27
mm3/frame | 0.093 (0.045) | 0.079 (0.035)
Statistical Analysis 1: Comparison: Arm 1: Prasugrel vs Arm 2: Placebo; Test type: Superiority; p = 0.97, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Arm 1: Prasugrel | Arm 2: Placebo
All-Cause Mortality (participants affected / at risk) | 2/42 | 1/42
Serious Adverse Events (participants affected / at risk) | 9/42 | 4/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Prasugrel (N=42) | Arm 2: Placebo (N=42)
Severe GUSTO bleeding (Blood and lymphatic system disorders) | 1 | 0
Death (General disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 2
Percutaneous Coronary Intervention (Cardiac disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT01560780/Prot_SAP_000.pdf